CLINICAL TRIAL: NCT03297281
Title: Multicenter Randomized Open-labelled Trial Which Aims to Show Non-inferiority of Adverse Events Risk During the Maintenance of Oral-anticoagulation in the Surgery of Benign Prostatic Hypertrophy by Laser Photovaporization
Brief Title: Stop or Ongoing Oral Anticoagulation in Patients Undergoing Pvp (SOAP)
Acronym: SOAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Vincent Misrai (Other)
Collaborators: Boston Scientific Corporation (Industry); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor-Investigator, Dr Vincent Misrai, Investigator coordinator, Clinique Pasteur
Organization: Clinique Pasteur (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-A01236-47
Record Dates: First submitted 2017-09-12; First posted 2017-09-29 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostatic Hyperplasia; Anticoagulant Adverse Reaction
Keywords: Photovaporization; Laser; Benign prostatic hyperplasia; Oral anticoagulation; Complication
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S1: maintenance (Experimental): Maintenance of OAC in surgery of BPH by PVP.
  Interventions: Other: Maintenance of OAC in surgery of BPH by PVP.
- S2 : discontinuation (Active Comparator): Discontinuation of OAC in surgery of BPH by PVP.
  Interventions: Other: Discontinuation of OAC in surgery of BPH by PVP.

INTERVENTIONS:
Other: Maintenance of OAC in surgery of BPH by PVP. — The maintenance of AVK or DOACs treatment in the perioperative setting (without interruption of oral treatment).
  Arms: S1: maintenance
Other: Discontinuation of OAC in surgery of BPH by PVP. — The discontinuation of AVK or DOACs treatment with perioperative heparin relay during postoperative course.
  Arms: S2 : discontinuation

SUMMARY:
Benign prostatic hyperplasia (BPH) is a very common pathology of the aging man with an incidence that rises from 40% in men aged 50 to 60 years to 90% in men over 80 years. Studies such as the MTOPS (the Medical Therapy of Prostatic Symptoms) study show that more than half of the patients recruited had an aggravation of their disease over time either by an increase in symptoms or by the appearance of complications such as acute retention of urine.

For benign symptomatic prostate hypertrophy, apart from any complication, first-line treatment is now a medical treatment. For patients who respond poorly to medical treatment or who have complications related to benign prostatic hypertrophy, the treatment becomes surgical. The reference treatment is endoscopic prostate resection (TURP). It is mainly to improve the safety of hemostasis in patients older and older and at significant surgical risk that new "minimally invasive" surgical techniques have emerged. Thus, lasers have been developed and are currently used as an alternative to the TURP. Used in clinical practice since 2000, prostatic photosensitive vaporization (PVP) relies on the absorption of a 532nm (green) wavelength laser beam by the oxyhemoglobin contained in richly vascularized prostate tissue.

Given the aging of the population, more and more patients are being treated with oral anticoagulants (Anti Vitamin K (AVK) or direct oral anticoagulants (DOACs)). Today there are about 1.4 million people on oral anticoagulants, 40% of whom are over 80 years of age. The peri-operative management of the AVK is currently based on the recommendations published by the FHA (French Health Authority) in 2008. Concerning the perioperative management of DOACs, the perioperative haemostasis interest group (GIHP) made proposals updated in September 2015.

Numerous studies published in the literature have concluded the feasibility of prostate removal surgery by PVP with greenlight laser without relay (or interruption) of AVK or DOACs because of the properties of hemostasis. But the levels of evidence for these studies remain low.

No study has focused on rigorously assessing the perioperative hemorrhagic risk associated with OAC therapy in patients eligible for PVP, and this is the originality of this study.

This study is a multicenter prospective randomized study whose objective is to show that the PVP performed in patients with OAC is not associated with an increase in perioperative hemorrhagic risk.

DETAILED DESCRIPTION:
SOAP is a non-inferiority, multicentric, open-labelled, two parallel arms study.

The expected benefits are to foster and make the perioperative management of OAC safer in patients undergoing BPH surgery with PVP.

ELIGIBILITY:
Inclusion Criteria:

* Prostate volume < or = 30 gr
* Micturition disorders resistant to medical treatment related to HBP and/or complications related to BPH (retention, lithiasis...)
* Patient candidate for photovaporization of the prostate
* Patient under treatment AVK (Anti Vitamin K) for more than 3 months with an objective of INR (International Normalized Ratio) between 2 and 3 or patient under DOACs (Direct Oral Anti-coagulants) for more than 3 months
* Unprotected major
* Patient affiliated to a social security scheme or equivalent
* Patient is willing and able to comply with all study requirements and to sign a study-specific informed consent form.

Exclusion Criteria:

* History of prostate cancer
* Previous pelvic radiotherapy
* History of stenosis of the urethra
* Patient with one or more bladder polyps
* Patient under antiplatelet agent other than aspirin
* Allergy to heparin or history of heparin-induced thrombocytopenia
* Patients under anticoagulant injectable therapy at baseline (heparin, LMWH (Low Molecular Weight Heparin), fondaparinux)
* Any mechanical prosthetic heart valve
* Stroke (ischemic or hemorrhagic), systemic embolism or transient ischemic attack within past 12 weeks
* Venous thromboembolism (deep vein thrombosis and/or pulmonary embolism) within past 12 weeks
* Major bleeding within past 6 weeks
* Severe renal insufficiency (calculated creatinine clearance < 30 mL / min)
* Thrombocytopenia (platelet count < 100 x 10^9 / L)
* Life expectancy < 1 month
* Condition that impairs compliance with trial protocol (e.g. cognitive impairment, uncontrolled psychiatric condition, geographic inaccessibility)
* Contra-indication to PVP surgery or contra-indication to general anesthesia
* Protected patients : majors under some form of guardianship
* Patient participating in another clinical study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with at least one complication classified higher or equal to grade 2 according to the Clavien classification related to maintenance of oral-anticoagulant (OAC) during the surgical resection of BPH by laser at 1 month | Between day 0 (day of the surgery) and day 30 (1 month after surgery)

SECONDARY OUTCOMES:
Number of patients with at least one hemorrhagic complication related to maintenance of oral-anticoagulant (OAC) during the surgical resection of BPH by laser at 1 month, 3 months and 6 months | At 1 month, 3 months and 6 months
  Haemorrhagic complications are defined by hematuria, bladder clotting removed from patient bed or operating room.
Number of patients with at least one thrombotic complication related to maintenance of oral-anticoagulant (OAC) during the surgical resection of BPH by laser at 1 month, 3 months and 6 months | At 1 month, 3 months and 6 months
  Thrombotic complications are defined by stroke, transient ischemic attacks and systemic embolisms.
Duration of hospitalization related to perioperative management of anticoagulants will be measured at the patient's discharge | At the patient's discharge, on average 3 days after surgery
Prostatic residual volume will be measured to evaluate the quality of resection under oral-anticoagulant at 1 month, 3 months, and 6 months | At 1 month, 3 months and 6 months
PSA level will be measured to evaluate the quality of resection under oral-anticoagulant at 1 month, 3 months, and 6 months | At 1 month, 3 months and 6 months
Questionnaires International Prostate Symptom Score (IPSS) will be complemented by patients to evaluate the functional success of surgery under oral-anticoagulant at 1 month, 3 months and 6 months | At 1 month, 3 months and 6 months
International Continence Society (ICS) will be complemented by patients to evaluate the functional success of surgery under oral-anticoagulant at 1 month, 3 months and 6 months | At 1 month, 3 months and 6 months
Volume of post-voiding residue will be measured to evaluate the functional success of surgery under oral-anticoagulant at 1 month, 3 months and 6 months | At 1 month, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Misrai, Dr, Principal Investigator — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan SA, McConnell JD, Roehrborn CG, Meehan AG, Lee MW, Noble WR, Kusek JW, Nyberg LM Jr; Medical Therapy of Prostatic Symptoms (MTOPS) Research Group. Combination therapy with doxazosin and finasteride for benign prostatic hyperplasia in patients with lower urinary tract symptoms and a baseline total prostate volume of 25 ml or greater. J Urol. 2006 Jan;175(1):217-20; discussion 220-1. doi: 10.1016/S0022-5347(05)00041-8. PMID 16406915
- [Background] Rosen R, Altwein J, Boyle P, Kirby RS, Lukacs B, Meuleman E, O'Leary MP, Puppo P, Robertson C, Giuliano F. Lower urinary tract symptoms and male sexual dysfunction: the multinational survey of the aging male (MSAM-7). Eur Urol. 2003 Dec;44(6):637-49. doi: 10.1016/j.eururo.2003.08.015. PMID 14644114
- [Background] Thomas JA, Tubaro A, Barber N, d'Ancona F, Muir G, Witzsch U, Grimm MO, Benejam J, Stolzenburg JU, Riddick A, Pahernik S, Roelink H, Ameye F, Saussine C, Bruyere F, Loidl W, Larner T, Gogoi NK, Hindley R, Muschter R, Thorpe A, Shrotri N, Graham S, Hamann M, Miller K, Schostak M, Capitan C, Knispel H, Bachmann A. A Multicenter Randomized Noninferiority Trial Comparing GreenLight-XPS Laser Vaporization of the Prostate and Transurethral Resection of the Prostate for the Treatment of Benign Prostatic Obstruction: Two-yr Outcomes of the GOLIATH Study. Eur Urol. 2016 Jan;69(1):94-102. doi: 10.1016/j.eururo.2015.07.054. Epub 2015 Aug 15. PMID 26283011
- [Background] Misrai V, Roupret M, Guillotreau J, Bordier B, Bruyere F. [Greenlight((R)) photoselective vaporisation for benign prostatic hyperplasia: a systematic review]. Prog Urol. 2013 Feb;23(2):77-87. doi: 10.1016/j.purol.2012.10.013. Epub 2012 Nov 26. French. PMID 23352299
- [Background] Peyronnet B, Cornu JN, Roupret M, Bruyere F, Misrai V. Trends in the Use of the GreenLight Laser in the Surgical Management of Benign Prostatic Obstruction in France Over the Past 10 Years. Eur Urol. 2015 Jun;67(6):1193-1195. doi: 10.1016/j.eururo.2015.01.003. Epub 2015 Jan 17. No abstract available. PMID 25605646
- [Background] Ruszat R, Wyler S, Forster T, Reich O, Stief CG, Gasser TC, Sulser T, Bachmann A. Safety and effectiveness of photoselective vaporization of the prostate (PVP) in patients on ongoing oral anticoagulation. Eur Urol. 2007 Apr;51(4):1031-8; discussion 1038-41. doi: 10.1016/j.eururo.2006.08.006. Epub 2006 Aug 18. PMID 16945475
- [Background] Reich O, Bachmann A, Siebels M, Hofstetter A, Stief CG, Sulser T. High power (80 W) potassium-titanyl-phosphate laser vaporization of the prostate in 66 high risk patients. J Urol. 2005 Jan;173(1):158-60. doi: 10.1097/01.ju.0000146631.14200.d4. PMID 15592063
- [Background] Charbonneau H, Pathak A, Albenque JP, Misrai V. Greenlight photovaporization of the prostate in patients under rivaroxaban: Lesson learned after the first cases. Prog Urol. 2016 Apr;26(5):273-5. doi: 10.1016/j.purol.2016.02.002. Epub 2016 Mar 9. No abstract available. PMID 26970929
- [Background] Douketis JD, Spyropoulos AC, Kaatz S, Becker RC, Caprini JA, Dunn AS, Garcia DA, Jacobson A, Jaffer AK, Kong DF, Schulman S, Turpie AG, Hasselblad V, Ortel TL; BRIDGE Investigators. Perioperative Bridging Anticoagulation in Patients with Atrial Fibrillation. N Engl J Med. 2015 Aug 27;373(9):823-33. doi: 10.1056/NEJMoa1501035. Epub 2015 Jun 22. PMID 26095867
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] Malek RS, Kuntzman RS, Barrett DM. High power potassium-titanyl-phosphate laser vaporization prostatectomy. J Urol. 2000 Jun;163(6):1730-3. PMID 10799170
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Bachmann A, Tubaro A, Barber N, d'Ancona F, Muir G, Witzsch U, Grimm MO, Benejam J, Stolzenburg JU, Riddick A, Pahernik S, Roelink H, Ameye F, Saussine C, Bruyere F, Loidl W, Larner T, Gogoi NK, Hindley R, Muschter R, Thorpe A, Shrotri N, Graham S, Hamann M, Miller K, Schostak M, Capitan C, Knispel H, Thomas JA. 180-W XPS GreenLight laser vaporisation versus transurethral resection of the prostate for the treatment of benign prostatic obstruction: 6-month safety and efficacy results of a European Multicentre Randomised Trial--the GOLIATH study. Eur Urol. 2014 May;65(5):931-42. doi: 10.1016/j.eururo.2013.10.040. Epub 2013 Nov 11. PMID 24331152
- [Background] Peyronnet B, Pradere B, Brichart N, Bodin T, Bertrand P; Members of French Group of GreenLight Users; Bruyere F. Complications associated with photoselective vaporization of the prostate: categorization by a panel of GreenLight users according to Clavien score and report of a single-center experience. Urology. 2014 Sep;84(3):657-64. doi: 10.1016/j.urology.2014.05.028. PMID 25168547
- [Derived] Charbonneau H, Pasquie M, Peyronnet B, Descazeaud A, Barry-Delongchamps N, Della Negra E, Mathieu R, Karsenty G, Long JA, Ballereau C, Azzouzi AR, Pradere B, Bruyere F, Fournier G, Lebdai S, Calves J, Corbel L, Vincendeau S, Fiard G, Thuillier C, Descotes JL, Colin P, Culty T, Hesbois A, Fuzier V, Savy N, Pathak A, Albaladejo P, Samama CM, Guerrero F, Misrai V. Stopping or maintaining oral anticoagulation in patients undergoing photoselective vaporization of the prostate (SOAP) surgery for benign prostate obstruction: study protocol for a multicentre randomized controlled trial. Trials. 2018 Dec 27;19(1):705. doi: 10.1186/s13063-018-3066-9. PMID 30587221
- See also: Access the 06/03/2017. — http://sfar.org/wp-content/uploads/2015/09/Reactualisation-GIHP_AOD_actes-programmes_Septembre-20151.pdf
- See also: Caroline Elie, Emmanuel Touze, Non-inferiority tests, Blood thrombosis vessels 24(2), pp.93-9, 2012. — http://www.jle.com/fr/revues/stv/e-docs/les_essais_de_non_inferiorite_292550/article.phtml